CLINICAL TRIAL: NCT06530784
Title: Cryoablation Combined With PD-1 Antibody and Bevacizumab for Hepatocellular Carcinoma After Progression of PD-1/L1 Antibody Treatment: a Pilot Clinical Study
Brief Title: Cryoablation Combined With PD-1 Antibody and Bevacizumab for Hepatocellular Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZS-IR-205R
Record Dates: First submitted 2024-07-22; First posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Carcinoma, Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Cryosurgery; Bevacizumab

STUDY DESIGN:
Intervention Model Description: Cryoablation combined with PD-1 antibody and bevacizumab
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment group (Experimental): Cryoablation combined with PD-1 antibody and bevacizumab
  Interventions: Procedure: Cryoablation; Drug: PD-1 antibody and bevacizumab

INTERVENTIONS:
Procedure: Cryoablation — After the completion of screening, the subjects received cryoablation treatment
Drug: PD-1 antibody and bevacizumab — Three days after cryoablation, the patients receive intravenous infusion of Tislelizumab (200mg, with 100mL of normal saline) and Bevacizumab (dose 15mg/kg, with 100mL of normal saline) .The patients will receive Tislelizumab (200 mg, with 100 mL of normal saline) and Bevacizumab (15 mg/kg, with 100 mL of normal saline) once every 3 weeks until disease progression.

SUMMARY:
To explore the safety and efficacy of cryoablation combined with PD-1 antibody and bevacizumab for patients with hepatocellular carcinoma resistance to PD-1/L1 antibody.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 80 years old, and expected survival is longer than 3 months
2. Clinically or pathologically diagnosed as primary hepatocellular carcinoma
3. Disease progression assessed according to mRECIST criteria after PD-1/L1 antibody treatment
4. Child-Pugh score of liver function A/B (< 7)
5. At least one lesion is suitable for mRECIST assessment
6. Strength score (ECOG): 0-1
7. The patient and/or family members agree to join the clinical trial and sign the informed consent form

Exclusion Criteria:

1. Patients whose tumor lesions are not suitable for ablation as assessed by the surgeon
2. Tumor burden greater than ≥70%, or tumor is not suitable for mRECIST standard evaluation
3. Patients with chronic viral hepatitis (hepatitis B, hepatitis C) have a viral load greater than 10^4 before receiving treatment or do not continue to take antiviral drugs regularly
4. Pregnant patients
5. Combined with other malignant tumors, or have a history of other malignant tumors within 3 years
6. Active autoimmune disease, confirmed immunodeficiency, history of systemic steroid medication
7. Severe renal dysfunction: creatinine (Cr) > 2 mg/dL or creatinine clearance (CCr) <30 mL/min, severe heart, lung, brain and other important organ diseases
8. History of gastrointestinal bleeding within 3 months
9. Unable to cooperate with ablation surgery
10. Severe gastroesophageal varices

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-07-31 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | Up to 2 years
  mRECIST is used as the evaluation criterion for CT/MRI imaging at each follow-up visit.

SECONDARY OUTCOMES:
Time to progress | Up to 2 years
  mRECIST is used as the evaluation criterion for CT/MRI imaging at each follow-up visit.
Objective Response Rate | Up to 2 years
  mRECIST is used as the evaluation criterion for CT/MRI imaging at each follow-up visit.
Overall survival | Up to 2 years
  According to medical documents or descriptions of the patient's family
Adverse events | Up to 2 years
  CTCAE v5.0 is used to assess adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Jian Zhou, Principal Investigator — Fudan University
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China